CLINICAL TRIAL: NCT01500902
Title: The Assessment of Novel Functional Risk Factors for the Prediction of Cardiovascular Events in Vulnerable Patients Following Acute Coronary Syndrome
Brief Title: Prediction of Cardiovascular Events in Vulnerable Patients Following Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Qatar National Research Fund (Other)
Responsible Party: Principal Investigator, Amir Lerman, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-000047
Record Dates: First submitted 2011-11-22; First posted 2011-12-29 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome (ACS); Percutaneous Intervention (PCI); Coronary Stent (CStent); Percutaneous Transluminal Coronary Angioplasty (PTCA); stent placement; balloon angioplasty
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vascular testing (Other): We are assessing vascular testing in patients presenting with acute coronary syndrome to determine if this type of testing will help identify which patients are more likely at risk to have another heart attack.
  Interventions: Other: EndoPAT testing (non invasive device); Other: WatchPAT testing (non-invasive device)

INTERVENTIONS:
Other: EndoPAT testing (non invasive device) — Using the EndoPAT device, we will assess endothelial function.
  Other Names: Itamar EndoPAT 2000
Other: WatchPAT testing (non-invasive device) — Using the WATCHPAT device we will assess sleep apnea.
  Other Names: Itamar WatchPAT 200

SUMMARY:
The purpose of this study is to determine if testing patients for endothelial dysfunction will help identify which patients are more likely at risk to have another heart attack in the future. Study participants will undergo mental stress testing while at the same time being connected to a device that measures endothelial function via the Endopat device. These same participants will also undergo a sleep study via the Watchpat device.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing revascularization by percutaneous intervention (PCI) for Acute Coronary Syndrome (ACS) at Mayo (STEMI and NonSTEMI patients)
2. Age greater than 18

Exclusion Criteria:

1. Patients likely not to complete the study due to co-morbid conditions (end stage renal disease; liver failure; malignancies)
2. Inability to sign a consent form or availability for follow up
3. Patients unable to tolerate the blood pressure cuff inflation on both arms
4. patients with tremors
5. sustained non-sinus cardiac arrhythmias
6. acrylic finger nails
7. permanent pacemaker
8. color blindness
9. use of alpha blockers and short acting nitrates < 3 hours before study
10. Federal Medical Center inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Unstable Angina, Myocardial Infarction, Repeat Revascularization, Cardiac Death, Stroke | Will determine with statistical analysis after all patients have had 2 year follow-up

SECONDARY OUTCOMES:
Quality of Life | 6 months post revascularization.
  Quality of Life as assessed by SF12

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States